CLINICAL TRIAL: NCT02049645
Title: The Suitability of Sniff Dog as a Tool in Screening Tumors-- a Prospective Observational Study
Brief Title: The Suitability of Sniff Dog as a Tool in Screening Tumors
Status: Recruiting | Type: Observational
Sponsor: Chang-Qing Gao (Other)
Responsible Party: Sponsor-Investigator, Chang-Qing Gao, MD PhD, Central South University
Organization: Central South University (Other)
Other Study IDs: Xiang-Ya 0001
Record Dates: First submitted 2014-01-25; First posted 2014-01-30 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Neoplasia
Keywords: lung cancer; breast cancer
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- faculty staff and their adult family members: faculties and their adult family members of the Third Xiang-Ya Hospital

SUMMARY:
Previous studies have demonstrated that sniff dogs can identify cancer patients from healthy subjects through sniffing exhaled breath air or blood or serum or urine or feces. It is hypothesized that sniff dogs may be used as a tool in screening cancer patients in health examination. Trained dogs will sniff serum from participants who are attending the annual health examination to identify potential or high risk subjects, and the results will be compared with the outcome of the traditional health examination, and the high risk subjects will be followed periodically for at least five years.

ELIGIBILITY:
Inclusion Criteria:

* old than 20 years
* currently without cancer diagnosed with pathological examination
* allow the study team to examine his/her case history and incoming record

Exclusion Criteria:

* cancer patients with pathological diagnosis
* who does not allow the study team to examine his/her case history and incoming record

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Third Xiang-Ya Hospital staff members and their adult family members who wish to participate the study.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2014-01; Primary Completion 2024-12-31 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity in screening cancer patients | up to 5 years
  The results that obtained from the dogs will be compared with these of the pathological examinations. Sensitivity = the No. of patients identified by the dogs as cancers / the No. of patients suffering from cancer confirmed by pathological examination. Specificity = No. of subjects signaled by the dog as non-cancers / No. of subjects confirmed by pathological examination or the currently used methods as non-cancer subjects or at the end of the study, 5 years later still without cancer.

SECONDARY OUTCOMES:
Behavior patterns of sniff dogs to different diseases | up to 5 years
  The behavior (lying before the tank for positive, neglecting the tanks) of the dog will be recorded and compared with the results of the pathological examination.

OTHER OUTCOMES:
The substances used by the sniff dogs to identifying tumors | up to 5 years
  GCMS etc will be used to compare the volatile compounds between the sera from cancers patients and the from normal subjects, the suspected VOCs will be tested by the dog for conformation.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Qing Gao, MD PhD, Principal Investigator — Central South University
Locations (1):
- The Third Xiang-Ya Hospital, Changsha, Hunan, China

REFERENCES:
- [Background] Ehmann R, Boedeker E, Friedrich U, Sagert J, Dippon J, Friedel G, Walles T. Canine scent detection in the diagnosis of lung cancer: revisiting a puzzling phenomenon. Eur Respir J. 2012 Mar;39(3):669-76. doi: 10.1183/09031936.00051711. Epub 2011 Aug 18. PMID 21852337
- [Background] Church J, Williams H. Another sniffer dog for the clinic? Lancet. 2001 Sep 15;358(9285):930. doi: 10.1016/S0140-6736(01)06065-2. No abstract available. PMID 11575380
- [Background] Willis CM, Church SM, Guest CM, Cook WA, McCarthy N, Bransbury AJ, Church MR, Church JC. Olfactory detection of human bladder cancer by dogs: proof of principle study. BMJ. 2004 Sep 25;329(7468):712. doi: 10.1136/bmj.329.7468.712. PMID 15388612
- [Background] McCulloch M, Jezierski T, Broffman M, Hubbard A, Turner K, Janecki T. Diagnostic accuracy of canine scent detection in early- and late-stage lung and breast cancers. Integr Cancer Ther. 2006 Mar;5(1):30-9. doi: 10.1177/1534735405285096. PMID 16484712
- [Background] Horvath G, Jarverud GA, Jarverud S, Horvath I. Human ovarian carcinomas detected by specific odor. Integr Cancer Ther. 2008 Jun;7(2):76-80. doi: 10.1177/1534735408319058. Epub 2008 May 27. PMID 18505901